CLINICAL TRIAL: NCT03758287
Title: A Phase Ib, Multi-center, Open Label Study of Ningetinib (CT053PTSA) in Combination With Gefitinib in Stage IIIB or IV NSCLC Patients With EGFR Mutation and T790M Negative Who Have Progressed After EGFR TKI Therapy
Brief Title: Ningetinib (CT053PTSA) Plus Gefitinib in Stage IIIB or IV NSCLC Patients With EGFR Mutation and T790M Negative
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DCT053-16-001
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT053PTSA +Gefitinib (Experimental): Patients will receive CT053PTSA and gefitinib over a 28-day cycle until progressive disease, intolerable toxicity or subject's withdrawal from treatment.
  CT053PTSA will be administered daily, at a dose of 30 mg/40mg/60mg orally .
  Gefitinib will be administered daily, at a dose of 250 mg orally .
  Interventions: Drug: CT053PTSA; Drug: Gefitinib

INTERVENTIONS:
Drug: CT053PTSA
  Other Names: Ningetinib
Drug: Gefitinib
  Other Names: Iressa

SUMMARY:
This is a phase Ib, multi-center, open label study evaluating the safety and efficacy of CT053PTSA in combination with gefitinib in patients with EGFR mutation, T790M negative NSCLC who have progressed after EGFR TKI treatment.

DETAILED DESCRIPTION:
This study is being carried out in two parts, part 1 and part 2.

Part 1: This is the dose-escalation part. The primary purpose of the part 1 portion is to determine the dose limiting toxicity (DLT) and maximum tolerated dose (MTD), and recommend the appropriate doses of CT053PTSA in combination with gefitinib for further studies.

Part 2: This is the expansion part. The part 2 portion of this study will continue to evaluate the safety and efficacy of the combination of CT053PTSA and gefitinib , at the appropriate doses recommended in Part 1, in patients with EGFR mutation, T790M negative NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Stage IIIB or IV NSCLC
* Resistance to EGFR TKI (1st, 2nd or 3rd generation)
* Histological or cytological evidence of EGFR mutation and T790M negative after progression on last EGFR TKI therapy
* c-Met GCN ≥ 6 or cluster amplification is required if participant is resistant to1st or 2nd generation EGFR-TKI ;c-MET GCN statue is not required, If participant is resistant to3rd generation EGFR-TKI （osimertinib）；
* Measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* Toxicity recovered to NCI CTCAE v.4.03 Grade ≤1 from previous treatments (except alopecia)
* ECOG performance status (PS) 0 or 1
* Life expectancy of ≥ 12 weeks
* Adequate organ function

Exclusion Criteria:

* Prior treatments

  * Chemotherapy, targeted therapy (except EGFR TKI), immunotherapy, radiotherapy, or major surgery within 4 weeks prior to study treatment
  * Nitrosourea and mitomycin chemotherapy within 6 weeks prior to study treatment
  * EGFR TKI treatment within 2 weeks prior to study treatment
  * Had received live vaccine within 4 weeks prior to study treatment
  * Had received any investigational agent from other clinical study within 4 weeks prior to study treatment or are currently participating in other clinical trials
  * Previous treatment with any other c-MET inhibitor or Axl inhibitor (eg, crizotinib, cabozantinib, volitinib, INC280)
* Symptomatic, untreated or unstable central nervous system metastases
* Spinal cord compression, carcinomatous meningitis or leptomeningeal diseaseonly (patient are only permitted if treated, asymptomatic and stable for at least 4 weeks prior to start of study treatment)
* Interstitial pneumonia or radiation pneumonitis
* Uncontrolled hypertension that require more than two anti-hypertensive agents to control, or systolic blood pressure (BP) >140mmHg or diastolic BP >90 mmHg before the first administration (BP is the mean blood pressure of two measures that 1 hours interval or above)
* Doppler ultrasound evaluation：Left ventricular ejection fraction < 50%
* Grade ≥ 2 of arrhythmia (assessed by NCI CTCAE 4.03), or symptomatic bradycardia, or male with QTCF > 450 ms or female with QTCF > 470 ms, or patients with a history of torsion or congenital QT prolonged syndrome long QT syndrome
* Certain factors that would preclude adequate absorption of CT053PTSA and gefitinib (eg. unable to swallow, chronic diarrhea, intestinal obstruction)
* Significant hemoptysis within 2 months prior to enrollment, or a daily hemoptysis volume is 2.5 ml or above
* Patients with evidence of bleeding tendency, including the following cases: gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ++ and above; or melena or hematemesis within 2 months; or visceral bleeding that may occur considered by investigator
* History of immunodeficiency, or other acquired or congenital immunodeficiency, or history of organ transplantation
* Any disease of the following bellowed within 12 months prior to administration: Myocardial infarction, severe angina, or unstable angina, coronary or peripheral artery bypass graft, congestive heart failure, or cerebrovascular events (including transient ischemic attack)
* Pulmonary embolism within 6 months prior to administration
* Active infection of hepatitis B, or infection of HIV
* Other malignancies within 5 years prior to enrollment, with the exception of carcinoma in situ of the cervix, basal or squamous cell skin cancer
* History of thyroid dysfunction, and the thyroid function cannot be maintained at the normal range with drugs.
* Serious electrolyte imbalance in the investigator's judgment
* Pregnant or lactating woman
* Any other reason the investigator considers the patient is not suitable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2023-07-17 (Estimated); Study Completion 2023-07-17 (Estimated)

PRIMARY OUTCOMES:
Part 1（dose-escalation part）: Maximum Tolerated Dose (MTD) | Cycle 1 Day 1 to Cycle 1 Day 28
  The maximum tolerated dose (MTD) of the CT053PTSA and gefitinib combination will be determined according to incidence of dose-limiting toxicity (DLT) assessed by NCI CTCAE v4.03
Part 2（expansion part）: Overall Response Rate | up to approximately 36 months
  Overall response rate (ORR), defined as a partial response (PR) or complete response (CR) occurring at any point post-treatment according to Response Evaluation Criteria in Solid Tumors as assessed by RECIST v1.1

SECONDARY OUTCOMES:
Number of patients with adverse events (AEs) as a measure of safety and tolerability | up to approximately 36 months
  Safety and tolerability will be assessed through AEs, via monitoring changes in physical examination, clinical laboratory parameters, vital signs and ECGs
Disease Control Rate (DCR) | up to approximately 36 months
  DCR, proportion of patients with best overall response of CR, PR or SD
Progression-free Survival (PFS) | up to approximately 36 months
  PFS, defined as time from date of treatment to disease progression or death due to any cause
Duration of Response (DOR) | up to approximately 36 months
  DOR, defined as time from the first documented CR or PR to first documented progression or death due to any cause
Overall Survival (OS) | up to approximately 60 months
  OS, defined as time from date of treatment to death due to any cause
Maximum observed plasma concentration (Cmax) | Cycle 1 Day1 and Day 28
  to assess the pharmacokinetic profile
Time of maximum observed plasma concentration (Tmax) | Cycle 1 Day1 and Day 28
  to assess the pharmacokinetic profile
Area under the plasma concentration time curve (AUC) | Cycle 1 Day1 and Day 28
  to assess the pharmacokinetic profile

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No